CLINICAL TRIAL: NCT06677567
Title: Comparison of the Efficacy of Self-Pressurizing Air-Q Intubation Laryngeal Airway and Proseal Laryngeal Mask in Elderly Patients
Brief Title: Air-Q and Proseal Laryngeal Mask in Elderly Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Zeynep Koc, principal investigator, Diskapi Yildirim Beyazit Education and Research Hospital
Other Study IDs: ZeynepKoc003
Record Dates: First submitted 2024-11-05; First posted 2024-11-06 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Postoperative Complications; Sore Throat
Keywords: Air-Q Laryngeal İntubating Airway; Oropharyngeal leak pressure; proseal larygeal mask; supraglottic airways
MeSH Terms: conditions — Postoperative Complications; Pharyngitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SP AİR Q group: under general anesthesia, patients inserted Air- Q intubating airway.
  Interventions: Other: Air-Q Intubating Airway
- Proseal Group: under general anesthesia, patients inserted proseal laryngeal mask.
  Interventions: Other: proseal laryngeal mask

INTERVENTIONS:
Other: Air-Q Intubating Airway — Patients will be inserted Air-Q Intubating Airway under general anesthesia
  Groups: SP AİR Q group
Other: proseal laryngeal mask — Patients will be inserted proseal laryngeal mask under general anesthesia.
  Groups: Proseal Group

SUMMARY:
Aged- related changes in upper airway anatomy may affect the overall performance of supraglottic airways significantly. In this study, investigator aim to compare the clinical performance, efficacy, and associated complications of the Proseal Laryngeal Mask and the Air-Q Intubation Laryngeal Airway in elderly patients.

DETAILED DESCRIPTION:
Elderly patients are vulnerable to perioperative pulmonary complications during intubation and extubation. Supraglottic airway devices (SADs) have been utilized as a relatively easy method of airway management for resuscitation and difficult intubations and are used during elective general anesthesia with reduced airway complications compared to endotracheal intubation. SADs may help maintain hemodynamic stability as they require less anesthetic agents compared to endotracheal intubation. With aging, parapharyngeal fat accumulation increases, leading to pharyngeal collapse in elderly patients. Additionally, structural changes in the respiratory tract combined with physiological alterations in respiration may reduce oxygen saturation, blunt the hypoxic response, and increase postoperative respiratory complications. Acquired changes in pharyngeal muscle activity with age are thought to increase the likelihood of bony structural changes, such as retrognathia, which is typically considered a difficult airway. Therefore, these age-related changes may impact the clinical performance of SADs. ProSeal LMA is one of the most commonly used supraglottic airway devices in clinical practice. It was developed by modifying the classic LMA in the 2000s and features an inflatable cuff. Additionally, it has a gastric channel for gastric aspiration adjacent to the airway tube. Recently, SGAs (supraglottic airways) that do not require manual cuff inflation have been increasingly used in various clinical situations due to the advantages of eliminating manual cuff inflation and monitoring cuff pressure. Air-Q connects to an airway tube via a communication port that allows self-regulation of cuff pressure in response to airway pressure. In this study, investigator aim to compare the clinical performance, efficacy, and associated complications of the Proseal Laryngeal Mask and the Air-Q Intubation Laryngeal Airway in elderly patients.

ELIGIBILITY:
Inclusion Criteria:

* 65-90 year-old patients
* American Society of Anesthesiologist Physical Status classification I-III,
* Undergoing an elective operation under general anesthesia in our hospital

Exclusion Criteria:

* Predicted difficult airway (Mallampati class 4, mouth opening < 3 cm, or thyromental distance < 6 cm)
* body mass index (BMI) > 40 kg/m2
* Patients with a high risk of aspiration (e.g., history of gastrectomy, -gastroesophageal reflux disease, or hiatal hernia),
* Unstable vital signs
* Cervical spine problems, Respiratory complications (e.g. recent pneumonia).

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged 65 to 90 years, both male and female, classified as ASA 1-3, will be included in the study if they undergo surgery with ProSeal LMA and Air-Q intubating airway.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-11-10 (Estimated); Primary Completion 2025-01-10 (Estimated); Study Completion 2025-01-20 (Estimated)

PRIMARY OUTCOMES:
Measurement of oropharyngeal leak pressure (OLP) | One minute after successful LMA placement
  One minute after successful LMA placement and fixation, oropharyngeal leak pressure (OLP) will be measured by setting the adjustable pressure limiting valve (APL) to 40 mmHg and maintaining a fresh gas flow of 3 L/min. The OLP will be recorded as the pressure at which an audible leak sound is heard from the mouth.

SECONDARY OUTCOMES:
SP Air-Q and proseal LMA insertion time | 3 minutes after induction of anesthesia
  Successful LMA placement will be confirmed by visualizing a square waveform on the ventilator and observing chest wall movement.

OTHER OUTCOMES:
ease of LMA placement | 3 minutes after induction of anesthesia
  he ease of LMA placement will be scored by the anesthesiologist on a scale from 1 to 4 (1: Successful on the first attempt with no resistance from the tissues; 2: Successful on the first attempt but with some tissue resistance during placement; 3: Moderate tissue resistance; 4: Failure to place the LMA).
maneuvers required for successful ventilation | 3 minutes after induction of anesthesia
  It will be recorded whether any further maneuvers are required: Gentle pushing or pulling of the LMA to adjust its depth, jaw-thrust maneuver, and flexion or extension of the head.
fiberoptic view grading | 3 minutes after induction of anesthesia
  The Brimacombe score will be used to evaluate the view obtained with fiberoptic bronchoscopy. 1: Vocal cords are not visible; 2: Vocal cords and anterior epiglottis are visible; 3: Vocal cords and posterior epiglottis are visible; 4: Vocal cords are visible.
Complications during SP_Air-Q and propseal LMA removal (emerge) | One minute after SP Air-Q removal
  Complications during SP_Air-Q and proseal LMA removal (emerge) such as breath-holding during emergence, airway obstruction, coughing, hypoxia (SpO2 < 90%), vomiting, lip-tongue-teeth trauma, and bleeding, will be recorded.
Sore throat | 1 hours postoperatively
  The presence or absence of sore throat will be recorded at the firsth postoperative hour.
Sore throat | 24 hours postoperatively
  The presence or absence of sore throat will be recorded at the 24th postoperative hour
dysphonia | 1 hours postoperatively
  The presence or absence of dysphonia will be recorded at the firsth postoperative hour
dysphonia | 24 hours postoperatively
  The presence or absence of dysphonia will be recorded at the 24th postoperative hour.

CONTACTS AND LOCATIONS:
Locations (1):
- Zeynep Koç, Yenimahalle, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim EM, Kim MS, Koo BN, Lee JR, Lee YS, Lee JH. Clinical efficacy of the classic laryngeal mask airway in elderly patients: a comparison with young adult patients. Korean J Anesthesiol. 2015 Dec;68(6):568-74. doi: 10.4097/kjae.2015.68.6.568. Epub 2015 Nov 25. PMID 26634080
- [Result] In CB, Cho SA, Lee SJ, Sung TY, Cho CK. Comparison of the clinical performance of airway management with the i-gel(R) and laryngeal mask airway SupremeTM in geriatric patients: a prospective and randomized study. Korean J Anesthesiol. 2019 Feb;72(1):39-46. doi: 10.4097/kja.d.18.00121. Epub 2018 Oct 22. PMID 30343563
- [Result] Lee JS, Kim DH, Choi SH, Ha SH, Kim S, Kim MS. Prospective, Randomized Comparison of the i-gel and the Self-Pressurized air-Q Intubating Laryngeal Airway in Elderly Anesthetized Patients. Anesth Analg. 2020 Feb;130(2):480-487. doi: 10.1213/ANE.0000000000003849. PMID 30320644
- [Result] Wahba RM, Ragaei MZ, Metry AA, Nakhla GM. Supraglottic Airway Devices for Elective Pediatric Anesthesia: I-gel versus Air-Q, Which is the Best? Anesth Essays Res. 2020 Jul-Sep;14(3):461-466. doi: 10.4103/aer.AER_107_20. Epub 2021 Mar 22. PMID 34092859